CLINICAL TRIAL: NCT02771756
Title: Randomized, Self Controlled Study on the Effect of Oral Supplement of Zhen Qi Shen Capsule Combined With Yu Yi Kang on Breast Cancer and Lung Cancer Patients With Chemotherapy
Brief Title: The Effect of Zhen Qi Shen Capsule Combined With Yu Yi Kang on Breast Cancer and Lung Cancer Patients With Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CH-BC-036
Record Dates: First submitted 2016-04-18; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer; Lung Cancer
Keywords: Breast cancer; Lung cancer; Nutritional support; Safety; Effectiveness
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms | interventions — Drug Therapy; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test group (Experimental): Zhen qishen capsule (2 capsules, Bid) and Oral Supplement of Yuyikang (50g, Bid), a total of 150 people, are used for 42 days continuously.
  Interventions: Dietary Supplement: zhen qishen capsule and Oral Supplement of Yuyikang; Radiation: chemotherapy; Other: nutrition education
- placebo group (Placebo Comparator): Zhen qishen capsule placebo (2 capsules, Bid) and Oral Supplement of Yuyikang placebo (50g,Bid), a total of 150 people, are used for 42 days continuously.
  Interventions: Dietary Supplement: zhen qishen capsule placebo and Oral Supplement of Yuyikang placebo; Radiation: chemotherapy; Other: nutrition education

INTERVENTIONS:
Dietary Supplement: zhen qishen capsule and Oral Supplement of Yuyikang
  Arms: test group
Dietary Supplement: zhen qishen capsule placebo and Oral Supplement of Yuyikang placebo
  Arms: placebo group
Radiation: chemotherapy
Other: nutrition education

SUMMARY:
The purpose of this study is to research more reasonable and safe methods of nutritional support to improve the nutritional status of tumor patients, which guarantees the anti-tumor treatment such as chemotherapy.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled clinical trials. 300 patients were randomly divided into 2 groups for its own control study.

Test group: Zhen qishen capsule (2 capsules, Bid) and Oral Supplement of Yuyikang (50g,Bid), a total of 150 people, are used for 42 days continuously.

Placebo group: Zhen qishen capsule placebo (2 capsules, Bid) and Oral Supplement of Yuyikang placebo (50g, Bid), a total of 150 people, are used for 42 days continuously.

The subjects were randomized to AB or BA parallely, and the two groups were given chemotherapy and nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years old
* Breast or lung cancer was diagnosed by pathology or cytology
* ECOG score: 0-2 points
* PG-SGA: 2-8 points, while the weight loss within 3 months less than 5%
* The organ function is good, with chemotherapy index. ANC is equal to or over 1.5 * 10^9/L, PLT is equal to or over 100* 10^9/L, HGB is equal to or over 90g/L
* Bilirubin is equal to or less than 1.5 times of the normal upper limit, AP, AST, ALT is less than or equal to 2 times of normal upper limit
* Ccr is equal to or over 50mL/min
* Life expectancy is equal to or over 12 weeks

Exclusion Criteria:

* Complete or incomplete intestinal obstruction
* A severe infection or difficult to control diabetes
* History of organ transplantation, or current use of immunosuppressive agents
* An intervention in nutritional supplements, or a metabolic disorder
* Parenteral nutrition must be applied
* Alcoholism or drug addiction
* Pregnancy or lactation, or women of childbearing age refuse contraception
* There are potential factors that interfere with the mental, psychological, family, social or geographical and other factors of the research project
* There are other diseases that may interfere with the results of this study, such as the second primary tumor
* For any other reason, the researchers were unable to complete the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Weight change rate | 6 weeks and 9 weeks after baseline.
Siderophilin change status | 6 weeks and 9 weeks after baseline.
Interleukin 1 change status | 6 weeks and 9 weeks after baseline.
interleukin 6 change status | 6 weeks and 9 weeks after baseline.
Tumor Necrosis Factor α change status | 6 weeks and 9 weeks after baseline.

SECONDARY OUTCOMES:
Change status of the Gripping Power | 6 weeks and 9 weeks after baseline.
Prealbumin Blood Examination change status | 6 weeks and 9 weeks after baseline.
Albumin change status | 6 weeks and 9 weeks after baseline.
Total Bilirubin change status | 6 weeks and 9 weeks after baseline.
Bilirubin Direct change status | 6 weeks and 9 weeks after baseline.
Indirect Bilirubin change status | 6 weeks and 9 weeks after baseline.
Alkaline Phosphatase change status | 6 weeks and 9 weeks after baseline.
Alanine Aminotransferase change status | 6 weeks and 9 weeks after baseline.
Aspartate Aminotransferase change status | 6 weeks and 9 weeks after baseline.
Serum Creatinine change status | 6 weeks and 9 weeks after baseline.
Urine Nitrogen change status | 6 weeks and 9 weeks after baseline.
Lymphocyte Number change status | 6 weeks and 9 weeks after baseline.
Hemoglobin change status | 6 weeks and 9 weeks after baseline.

OTHER OUTCOMES:
Quality of life questionnaire(QOL-C30) | At baseline,6 weeks and 9 weeks after baseline.
Scored Patient-Generated Subjective Global Assessment(PG-SGA) | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, MD, Principal Investigator — Chief physician
Locations (1):
- National Cancer Institute, Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes